CLINICAL TRIAL: NCT05297305
Title: Onlay Versus Inlay Humeral Component in Reverse Total Shoulder Arthroplasty: A Prospective, Randomized Trial
Brief Title: Onlay Versus Inlay Humeral Component in Reverse Total Shoulder Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding limitations and slow enrollment
Sponsor: Corewell Health East (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Dr. Alex Martusiewicz, staff physician, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-000
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Arthritis Shoulder; Rotator Cuff Injuries
Keywords: shoulder function; shoulder pain; shoulder range of motion
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomized double-blind trial of two active comparators.
Who Masked: Participant, Outcomes Assessor
Masking Description: Key personnel not collecting data will perform randomization and inform surgeon of the group assignment, keeping data collection blinded. The participant will also remain blinded to their assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Onlay Component-Tornier Ascend Flex stem (Active Comparator): Reverse Total Shoulder Arthroplasty using onlay component (tray placed at top of humerus)
  Interventions: Device: Tornier Ascend Flex stem
- Inlay Component-Tornier Perform Stem Reverse+ (Active Comparator): Reverse Total Shoulder Arthroplasty using inlay component (tray placed in humerus)
  Interventions: Device: Tornier Perform Stem Reverse+

INTERVENTIONS:
Device: Tornier Ascend Flex stem — Reverse Total Shoulder Arthroplasty using onlay component (tray placed at top of humerus)
  Arms: Onlay Component-Tornier Ascend Flex stem
Device: Tornier Perform Stem Reverse+ — Reverse Total Shoulder Arthroplasty using inlay component (tray placed in humerus)
  Arms: Inlay Component-Tornier Perform Stem Reverse+

SUMMARY:
The goal of this study is to compare the effect of different ways to place the component that goes at the top of the humerus (upper arm) in reverse total shoulder replacement. Some surgeons place the humeral tray component sitting on the bone while others place it in the bone. Changing the way that the humeral component is placed may change how much the arm can raise up or turn out/in after surgery for some patients. This study compares patients with inlay humeral component (tray sits in the upper arm bone) versus onlay humeral component (tray sits on top of the upper arm bone) to see if there are differences in range of motion or function after surgery.

DETAILED DESCRIPTION:
This study aims to determine if active external rotation two years postoperatively varies based on whether an inlay or onlay humeral component is used in reverse shoulder arthroplasty (RTSA). The study also aims to determine whether active forward elevation, abduction, scapular notching, and functional outcomes two years postoperatively vary based on whether an inlay or onlay humeral component is used in reverse shoulder arthroplasty. Patients undergoing primary RTSA by Dr. J. Michael Wiater, Dr. Brett Wiater, or Dr. Alexander Martusiewicz at Beaumont Health will be screened for eligibility. Following informed consent, participants will be randomised (1:1) to one of the following groups: 1) RTSA with inlay humeral component (Tornier Perform Stem Reverse+) or 2) RTSA with onlay humeral component (Tornier Ascend Flex stem). At baseline, participants will complete study questionnaires, receive a range-of-motion (ROM) exam, and standard of care x-rays and computed tomography (CT) scans. These evaluations will be repeated at 3 months, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary reverse total shoulder arthroplasty with the following components:

  1. Onlay group: Ascend Flex stem, Perform Reversed standard +3 lateralized 25mm baseplate with standard 36 mm glenosphere or +6 lateralized 25mm baseplate with 39mm glenosphere
  2. Inlay group: Perform Stem Reverse, Perform Reversed +3 lateralized 25mm baseplate with standard 36mm glenosphere or +6 lateralized 25mm baseplate with 39mm glenosphere
* Diagnosis of cuff tear arthropathy, massive cuff tear, or primary osteoarthritis with cuff tear
* Negative external rotation lag sign, ability to externally rotate beyond neutral
* Age 18 years or older

Exclusion Criteria:

* Revision arthroplasty
* Prior open shoulder surgery
* Concomitant tendon transfer (Latissimus Dorsi, Pectoralis Tendon, Lower Trapezius)
* Diagnosis of rheumatoid arthritis, infection, acute trauma or instability
* Patients not willing to undergo a standardized physical therapy protocol or home therapy program after surgical intervention
* Patient anatomy does not accommodate the study implants per surgeon discretion
* Pregnant, patient-reported
* Minors (under 18 years of age)
* Cognitively impaired based on a diagnosis of dementia, psychiatric disorder, or any cognitive deficit that will not allow for proper informed consent or answering of study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Active external rotation, 2 years | 2 years postoperative
  Range of motion of repaired shoulder, active external rotation. Measured with goniometer in degrees.

SECONDARY OUTCOMES:
Active external rotation, 3 months | 3 months postoperative
  Range of motion of repaired shoulder, active external rotation. Measured with goniometer in degrees.
Active external rotation, 1 year | 1 year postoperative
  Range of motion of repaired shoulder, active external rotation. Measured with goniometer in degrees.
Strength during active external rotation, 3 months | 3 months postoperative
  Strength measurement during active external rotation of repaired shoulder. Measured with dynamometer in pounds.
Strength during active external rotation, 1 year | 1 year postoperative
  Strength measurement during active external rotation of repaired shoulder. Measured with dynamometer in pounds.
Strength during active external rotation, 2 years | 2 years postoperative
  Strength measurement during active external rotation of repaired shoulder. Measured with dynamometer in pounds
Active forward elevation, 3 months | 3 months postoperative
  Range of motion of repaired shoulder, active forward elevation. Measured with goniometer in degrees.
Active forward elevation, 1 year | 1 year postoperative
  Range of motion of repaired shoulder, active forward elevation. Measured with goniometer in degrees.
Active forward elevation, 2 years | 2 years postoperative
  Range of motion of repaired shoulder, active forward elevation. Measured with goniometer in degrees.
Strength during active forward elevation, 3 months | 3 months postoperative
  Strength measured during active forward elevation of repaired shoulder. Measured with dynamometer in pounds.
Strength during active forward elevation, 1 year | 1 year postoperative
  Strength measured during active forward elevation of repaired shoulder. Measured with dynamometer in pounds.
Strength during active forward elevation, 2 years | 2 years postoperative
  Strength measured during active forward elevation of repaired shoulder. Measured with dynamometer in pounds.
Abduction, 3 months | 3 months postoperative
  Range of motion of repaired shoulder, abduction. Measured with goniometer in degrees.
Abduction, 1 year | 1 year postoperative
  Range of motion of repaired shoulder, abduction. Measured with goniometer in degrees.
Abduction, 2 years | 2 years postoperative
  Range of motion of repaired shoulder, abduction. Measured with goniometer in degrees.
Strength during abduction, 3 months | 3 months postoperative
  Strength measured during abduction of repaired shoulder. Measured with dynamometer in pounds.
Strength during abduction, 1 year | 1 year postoperative
  Strength measured during abduction of repaired shoulder. Measured with dynamometer in pounds.
Strength during abduction, 2 years | 2 years postoperative
  Strength measured during abduction of repaired shoulder. Measured with dynamometer in pounds.
Internal rotation, 3 months | 3 months postoperative
  Range of motion of repaired shoulder, internal rotation. Measured with goniometer in degrees.
Internal rotation, 1 year | 1 year postoperative
  Range of motion of repaired shoulder, internal rotation. Measured with goniometer in degrees.
Internal rotation, 2 years | 2 years postoperative
  Range of motion of repaired shoulder, internal rotation. Measured with goniometer in degrees.
Strength during Internal rotation, 3 months | 3 months postoperative
  Strength measured during internal rotation of repaired shoulder. Measured with dynamometer in pounds.
Strength during Internal rotation, 1 year | 1 year postoperative
  Strength measured during internal rotation of repaired shoulder. Measured with dynamometer in pounds.
Strength during Internal rotation, 2 years | 2 years postoperative
  Strength measured during internal rotation of repaired shoulder. Measured with dynamometer in pounds.
External rotation lag sign test, 3 months | 3 months postoperative
  Number of patients with positive external rotation lag sign test. The test is performed with the elbow passively flexed and repaired shoulder abducted 90 degrees by the examiner. Next, the examiner passively takes the patient's shoulder into a position of maximal external rotation. The patient is then instructed to hold that position. A positive test is if the patient cannot maintain the position and the shoulder rotates internally. A positive test indicates supraspinatus and infraspinatus tendon weakness.
External rotation lag sign test, 1 year | 1 year postoperative
  Number of patients with positive external rotation lag sign test. The test is performed with the elbow passively flexed and repaired shoulder abducted 90 degrees by the examiner. Next, the examiner passively takes the patient's shoulder into a position of maximal external rotation. The patient is then instructed to hold that position. A positive test is if the patient cannot maintain the position and the shoulder rotates internally. A positive test indicates supraspinatus and infraspinatus tendon weakness.
External rotation lag sign test, 2 years | 2 years postoperative
  Number of patients with positive external rotation lag sign test. The test is performed with the elbow passively flexed and repaired shoulder abducted 90 degrees by the examiner. Next, the examiner passively takes the patient's shoulder into a position of maximal external rotation. The patient is then instructed to hold that position. A positive test is if the patient cannot maintain the position and the shoulder rotates internally A positive test indicates supraspinatus and infraspinatus tendon weakness.
Drop arm test, 3 months | 3 months postoperative
  Number of patients with positive drop arm test of repaired shoulder, performed by passively abducting the patient's shoulder and observing for arm drop as the patient slowly lowers the arm to the waist. A positive test indicates supraspinatus dysfunction.
Drop arm test, 1 year | 1 year postoperative
  Number of patients with positive drop arm test of repaired shoulder, performed by passively abducting the patient's shoulder and observing for arm drop as the patient slowly lowers the arm to the waist. A positive test indicates supraspinatus dysfunction.
Drop arm test, 2 years | 2 years postoperative
  Number of patients with positive drop arm test of repaired shoulder, performed by passively abducting the patient's shoulder and observing for arm drop as the patient slowly lowers the arm to the waist. A positive test indicates supraspinatus dysfunction.
Lift off test, 3 months | 3 months postoperative
  Number of patients with positive lift off test. The test is performed by the patient performing internal rotation of repaired shoulder, by lifting the hand off the back while the examiner places pressure on the hand. The test is considered to be positive if the patient cannot resist, lift the hand off the back or if the patient compensates by extending the elbow and shoulder. A positive test indicates subscapularis weakness.
Lift off test, 1 year | 1 year postoperative
  Number of patients with positive lift off test. The test is performed by the patient performing internal rotation of repaired shoulder, by lifting the hand off the back while the examiner places pressure on the hand. The test is considered to be positive if the patient cannot resist, lift the hand off the back or if the patient compensates by extending the elbow and shoulder. A positive test indicates subscapularis weakness.
Lift off test, 2 years | 2 years postoperative
  Number of patients with positive lift off test. The test is performed by the patient performing internal rotation of repaired shoulder, by lifting the hand off the back while the examiner places pressure on the hand. The test is considered to be positive if the patient cannot resist, lift the hand off the back or if the patient compensates by extending the elbow and shoulder. A positive test indicates subscapularis weakness.
Belly press test, 3 months | 3 months postoperative
  Number of patients with positive belly press test. The patient is asked to press the palm of the hand against the abdomen and bring the elbow forward. The test is positive if the patient is unable to maintain maximal internal rotation of repaired shoulder, demonstrates weakness or the elbow deviates posteriorly. A positive test indicates subscapularis muscle dysfunction.
Belly press test, 1 year | 1 year postoperative
  Number of patients with positive belly press test. The patient is asked to press the palm of the hand against the abdomen and bring the elbow forward. The test is positive if the patient is unable to maintain maximal internal rotation of repaired shoulder, demonstrates weakness or the elbow deviates posteriorly. A positive test indicates subscapularis muscle dysfunction.
Belly press test, 2 years | 2 years postoperative
  Number of patients with positive belly press test. The patient is asked to press the palm of the hand against the abdomen and bring the elbow forward. The test is positive if the patient is unable to maintain maximal internal rotation of repaired shoulder, demonstrates weakness or the elbow deviates posteriorly. A positive test indicates subscapularis muscle dysfunction.
Functional impairment by American Shoulder and Elbow Surgeons' score (ASES), 3 months | 3 months postoperative
  Patients will complete a questionnaire of the repaired shoulder function and pain, with 100 maximum points. A score of 0 indicates no impairment (best outcome), and 100 indicates maximum impairment (worst outcome).
Functional impairment by American Shoulder and Elbow Surgeons' score (ASES), 1 year | 1 year postoperative
  Patients will complete a questionnaire of the repaired shoulder function and pain, with 100 maximum points. A score of 0 indicates no impairment (best outcome), and 100 indicates maximum impairment (worst outcome).
Functional impairment by American Shoulder and Elbow Surgeons' score (ASES), 2 years | 2 years postoperative
  Patients will complete a questionnaire of shoulder function and pain, with 100 maximum points. A score of 0 indicates no impairment (best outcome), and 100 indicates maximum impairment (worst outcome).
Quality of life by Western Ontario Osteoarthritis of the Shoulder score (WOOS), 3 months | 3 months postoperative
  Patients complete a questionnaire comprising 4 domains of: physical symptoms; sports, recreation and work; lifestyle; and emotions. Each question is answered using a visual analog scale with a possible score ranging from 0 to 100. There are 19 questions, and the total score ranges from 0 to 1900. A score of 1900 signifies that the patient has an extreme decrease in the shoulder-related quality of life (worst outcome), whereas a score of 0 signifies that the patient has no decrease in shoulder-related quality of life (best outcome).
Quality of life by Western Ontario Osteoarthritis of the Shoulder score (WOOS), 1 year | 1 year postoperative
  Patients complete a questionnaire comprising 4 domains of: physical symptoms; sports, recreation and work; lifestyle; and emotions. Each question is answered using a visual analog scale with a possible score ranging from 0 to 100. There are 19 questions, and the total score ranges from 0 to 1900. A score of 1900 signifies that the patient has an extreme decrease in the shoulder-related quality of life (worst outcome), whereas a score of 0 signifies that the patient has no decrease in shoulder-related quality of life (best outcome).
Quality of life by Western Ontario Osteoarthritis of the Shoulder score (WOOS), 2 years | 2 years postoperative
  Patients complete a questionnaire comprising 4 domains of: physical symptoms; sports, recreation and work; lifestyle; and emotions. Each question is answered using a visual analog scale with a possible score ranging from 0 to 100. There are 19 questions, and the total score ranges from 0 to 1900. A score of 1900 signifies that the patient has an extreme decrease in the shoulder-related quality of life (worst outcome), whereas a score of 0 signifies that the patient has no decrease in shoulder-related quality of life (best outcome).
Global Health, by Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) score, 3 months | 3 months postoperative
  Patients will complete the PROMIS-10 assessment of global health for the previous 7 days, a 10-question assessment where each statement is scored from 1 (poor health) to 5 (excellent health) on a Likert scale. A total score is summed from the 10 questions, resulting in a minimum of 10 and maximum of 50 points. Higher scores indicate better health (best outcome).
Global Health, by Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) score, 1 year | 1 year postoperative
  Patients will complete the PROMIS-10 assessment of global health for the previous 7 days, a 10-question assessment where each statement is scored from 1 (poor health) to 5 (excellent health) on a Likert scale. A total score is summed from the 10 questions, resulting in a minimum of 10 and maximum of 50 points. Higher scores indicate better health (best outcome).
Global Health, by Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) score, 2 years | 2 years postoperative
  Patients will complete the PROMIS-10 assessment of global health for the previous 7 days, a 10-question assessment where each statement is scored from 1 (poor health) to 5 (excellent health) on a Likert scale. A total score is summed from the 10 questions, resulting in a minimum of 10 and maximum of 50 points. Higher scores indicate better health (best outcome).
Visual Analog Scale measure of pain, 3 months | 3 months postoperative
  Shoulder-related pain reported by the patient for the repaired shoulder as a score on a visual analog scale from 0 to 10, where 0=no pain at all (best outcome), and 10=pain as bad as it can be (worst outcome).
Visual Analog Scale measure of pain, 1 year | 1 year postoperative
  Shoulder-related pain reported by the patient for the repaired shoulder as a score on a visual analog scale from 0 to 10, where 0=no pain at all (best outcome), and 10=pain as bad as it can be (worst outcome).
Visual Analog Scale measure of pain, 2 years | 2 years postoperative
  Shoulder-related pain reported by the patient for the repaired shoulder as a score on a visual analog scale from 0 to 10, where 0=no pain at all (best outcome), and 10=pain as bad as it can be (worst outcome).
Scapular notching, 3 months | 3 months postoperative
  Scapular notching of the repaired shoulder. Measured from radiographic evaluation and scored on the Sirveaux classification scale as Grade 1-4, where grade 1 indicates a defect that only involves the inferior pillar of the scapular neck (best outcome). In Grade 2, the notch contacts the lower screw. In Grade 3, erosion of the bone extends over the lower screw. In Grade 4, the notch extends under the baseplate (worst outcome).
Scapular notching, 1 year | 1 year postoperative
  Scapular notching of the repaired shoulder. Measured from radiographic evaluation and scored on the Sirveaux classification scale as Grade 1-4, where grade 1 indicates a defect that only involves the inferior pillar of the scapular neck (best outcome). In Grade 2, the notch contacts the lower screw. In Grade 3, erosion of the bone extends over the lower screw. In Grade 4, the notch extends under the baseplate (worst outcome).
Scapular notching, 2 years | 2 years postoperative
  Scapular notching of the repaired shoulder. Measured from radiographic evaluation and scored on the Sirveaux classification scale as Grade 1-4, where grade 1 indicates a defect that only involves the inferior pillar of the scapular neck (best outcome). In Grade 2, the notch contacts the lower screw. In Grade 3, erosion of the bone extends over the lower screw. In Grade 4, the notch extends under the baseplate (worst outcome).
Reoperation | 2 years postoperative
  Number of patients requiring reoperation of the same shoulder within 2 years.
Study-related adverse events | 2 years postoperative
  All adverse events determined by the PI to be probably or definitely related to study interventions (surgery or device).

CONTACTS AND LOCATIONS:
Overall Officials: Alex Martusiewicz, MD, Principal Investigator — Beaumont Health
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No